CLINICAL TRIAL: NCT06105827
Title: A Multicenter, Prospective, Randomized, Controlled Clinical Study of Ningmitai Capsule to Promote the Passage of Residual Fragments After Ureteroscopic Lithotripsy
Brief Title: Clinical Study of Ningmitai Capsule on Promoting the Passage of Residual Fragments After Ureteroscopic Lithotripsy
Acronym: 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMT16049S
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Ureteral Calculi
Keywords: Ureteral calculi; Lithotripsy of ureteral calculi; Ningmitai capsule; Residual fragments
MeSH Terms: conditions — Ureteral Calculi | interventions — Control Groups; Diclofenac; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Give antibiotics or diclofenac sodium suppository as needed.
  Interventions: Drug: Control group
- Ningmitai capsule (Experimental): Ningmitai Capsule (produced by Guiyang Xintian Pharmaceutical Co., Ltd.), 0.38 g/capsule, 4 capsules each time, 3 times a day. Course of treatment: 12 weeks
  Interventions: Drug: Ningmitai capsule
- Combined group (Ningmitai plus tamsulosin) (Experimental): Tamsulosin capsules, 0.2 mg/capsule, one capsule each time, once a day, were taken on the basis of Ningmitai group. Course of treatment: 12 weeks
  Interventions: Drug: Combined group (Ningmitai plus tamsulosin)

INTERVENTIONS:
Drug: Control group — Give antibiotics or diclofenac sodium suppository as needed.
  Other Names: diclofenac sodium
  Arms: Control group
Drug: Ningmitai capsule — Oral Ningmitai Capsule (produced by Guiyang Xintian Pharmaceutical Co., Ltd.), 0.38 g/capsule, 4 capsules each time, 3 times a day for 12 Weeks.
  Arms: Ningmitai capsule
Drug: Combined group (Ningmitai plus tamsulosin) — Tamsulosin capsules, 0.2 mg/capsule, one capsule each time, once a day, were taken on the basis of Ningmitai group for 12 Weeks.
  Other Names: Ningmitai plus tamsulosin
  Arms: Combined group (Ningmitai plus tamsulosin)

SUMMARY:
Objective: To observe the effect of Ningmitai capsule on ureteral calculi after lithotripsy and evaluate the safety of treatment.

Study Design: A multicenter, prospective, randomized, controlled clinical study design was adopted

Interventions:

control group: Give antibiotics or diclofenac sodium suppository as needed. Ningmitai group: Oral Ningmitai Capsule (produced by Guiyang Xintian Pharmaceutical Co., Ltd.), 0.38 g/capsule, 4 capsules each time, 3 times a day.

combination group (Ningmitai plus tamsulosin).: Tamsulosin capsules, 0.2 mg/capsule, one capsule each time, once a day, were taken on the basis of Ningmitai group.

DETAILED DESCRIPTION:
Sample size: 230

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as upper urinary calculi by B-ultrasound, kidney and upper bladder (KUB), intravenous urogram (IVU) or computerized tomography (CT) before surgery with the ages between 20 and 70 years.
2. Having ureteral residual fragments post URL and the diameter more than 5mm.
3. The lithotripsy went smoothly with expected outcomes and without any ureteral perforation, mucous exfoliation, kidney or bladder injury, serious bleeding or any other complications.
4. Willing and able to participate in this study and comply with all scheduled visits, treatment plans and complete the clinical observations.

Exclusion Criteria:

1. Pregnancy, severe diabetes, or renal insufficiency.
2. Ureteral stricture and lower urinary tract obstruction.
3. Concomitant treatment with α1-receptor antagonists, or Chinese traditional medicines who can be used to relieve stranguria and expel stone, or any other treatment that might interference the efficacy evaluation.
4. Unwilling or unable to comply with the administration regimen described in the protocol, or having an incomplete profile, hence their efficacy and safety couldn't be evaluated.
5. Severe adverse events and need to withdraw from the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
the stone expulsion time, stone-free time | From baseline to 12 weeks of treatment
  The diminishing or vanishing of residual fragment identified by post-surgery B-ultrasound or KUB could suggest a residual fragment expulsion. Evaluation with KUB showing the shadow of calculi disappearing completely followed by a confirmation using CT could suggest a residual fragment clearance.

SECONDARY OUTCOMES:
the stone expulsion rate and stone-free rate. | From baseline to 12 weeks of treatment
  The diminishing or vanishing of residual fragment identified by post-surgery B-ultrasound or KUB could suggest a residual fragment expulsion. Evaluation with KUB showing the shadow of calculi disappearing completely followed by a confirmation using CT could suggest a residual fragment clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Jingdong, Doctor, Principal Investigator — Wuhan First Hospital

IPD SHARING:
Plan to Share IPD: No